CLINICAL TRIAL: NCT04064697
Title: Impact of Anti-cytomegalovirus (Valganciclovir) Treatment in the Management of Relapsing Ulcerative Colitis (UC) Requiring Vedolizumab Therapy: a Randomized Clinical Trial Comparing a Strategy With or Without Antiviral Therapy.
Brief Title: Impact of Anti-cytomegalovirus Treatment in the Management of Relapsing Ulcerative Colitis Requiring Vedolizumab Therapy
Acronym: CYTOVEDO
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: low of inclusions
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18PH192; 2019-001032-54 (EudraCT Number)
Record Dates: First submitted 2019-08-20; First posted 2019-08-22 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2023-06

CONDITIONS: Ulcerative Colitis, Unspecified
Keywords: Ulcerative Colitis (UC); CytoMegaloVirus (CMV); Vedolizumab; Valganciclovir; Anti-TNF; Mayo score
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Valganciclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Patient will be treated by vedolizumab the standard of care alone.
- Experimental group (Experimental): Patient will be treated by vedolizumab the standard of care associated at valganciclovir.
  Interventions: Drug: Valganciclovir

INTERVENTIONS:
Drug: Valganciclovir — The experimental intervention consists of taking the treatment Valganciclovir 900 mg morning and evening for 3 weeks
  Other Names: antiviral therapy
  Arms: Experimental group

SUMMARY:
Ulcerative Colitis (UC) is an inflammatory bowel disease that can require the use of anti-TNF alpha therapy. When anti-TNF alpha failed to obtain a clinical response, the use of a new anti-integrin therapy, vedolizumab, can be proposed. The efficacy of vedolizumab has been assessed in a phase 3 study (GEMINI I), with response rates of 41.1% with vedolizumab vs 25.5% with placebo.

CytoMegaloVirus (CMV) reactivation has been associated with resistance to steroid and to several lines of immunosuppressive therapy. Antiviral therapy was proven to decrease the tissue viral load and to restore the response to immunosuppressive therapies (up to 80% in small group of patients). A recent meta-analysis supports the use of valganciclovir in case of CytoMegaloVirus (CMV) reactivation in active Ulcerative Colitis (UC).

Moreover, a study showed that the risk of CMV reactivation seems to be more important with vedolizumab than with anti TNF, and the risk of colectomy is higher in case of CytoMegaloVirus (CMV) reactivation (p<0.05).

DETAILED DESCRIPTION:
The hypothesis of this study is in Ulcerative Colitis (UC) patients with tissue CytoMegaloVirus (CMV) reactivation ; not responding to anti-TNF or without anti-TNF ; a treatment with valganciclovir, added to vedolizumab, could improve the clinical response.

ELIGIBILITY:
Inclusion Criteria:

* Patient with moderate to severe active Ulcerative Colitis (UC) defined by a Mayo score greater than 5
* Patient with an inflammatory outbreak of Ulcerative Colitis (UC) :

  * without anti-TNF
  * under anti-TNF (infliximab, adalimumab, golimumab) after induction (no primary response) or clinical recurrence (secondary failure).
* Having rectosigmoidoscopy with an endoscopic Mayo score≥ 2 with 2 biopsies of the inflammatory tissue
* Presence of a CytoMegaloVirus (CMV) infection in the inflammatory tissue (viral load greater than 5 IU / 100000 cells by qPCR)
* Patient with a negative pre-treatment assessment including HIV, HBV, HCV, HCV serology, a negative quantiferon or a history of tuberculosis preventive treatment adapted by Rifinah or Rimifon
* Signed informed consent

Exclusion Criteria:

* Patient with severe acute colitis
* Patient treated by ciclosporin or Prograf
* Patient with Human Immunodeficiency Virus (HIV)+, hepatitis B, hepatitis C, tuberculosis
* Clostridium difficile infection.
* Patient with intolerance or contraindications to current therapy
* Pregnant or starts breastfeeding
* Patient who received a live vaccine in the month preceding the study
* Patients with severe renal insufficiency defined by creatinine clearance <30ml/minute, or hemodialysed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2023-11-23 (Actual); Study Completion 2024-02-08 (Actual)

PRIMARY OUTCOMES:
Clinical response | Weeks 6
  Percentage of patients in clinical response. the clinical response is defined by the decrease in the total Mayo Score compared to the inclusion of at least 3 points and at least 30% with a decrease in the score of bleeding (item 2 of the Mayo sub-score) from at least one point or sub-score of bleeding from 0 or 1 point with or without anti-CMV treatment. The Mayo score includes 3 items: stool frequency, presence of blood in the stool, and overall assessment of the disease.

SECONDARY OUTCOMES:
Clinical remission | Weeks 6
  Percentage of patients in clinical remission defined by a total Mayo score <3 with an endoscopic score <2 and no clinical sub-score> 2.
Mucosal healing | Weeks 6
  Percentage of patients in mucosal healing defined by endoscopic mayo score <2
Viral load CytoMegaloVirus (CMV) | Weeks 6
  Value of viral load CytoMegaloVirus (CMV) by qPCR on inflammatory tissue in IU / 100000 cells.
clinical remission | Weeks 52
  Percentage of patients in clinical remission defined by a total Mayo score <3 with an endoscopic score <2 and no clinical sub-score> 2.
Rate of colectomy | Weeks 52
  Percentage of patients who required colectomy
Adverse effects | Weeks 52
  Number and severity of adverse effects
viral load of the Torque teno virus | Week 6
  performed on the blood tube and tissue biopsies

CONTACTS AND LOCATIONS:
Overall Officials: Pauline VEYRARD, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (8):
- France (8):
  - CH d'Annecy, Annecy
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CHU de Lyon Sud, Lyon
  - CHU de Montpellier, Montpellier
  - CHU de Nice, Nice
  - APHP - Hôpital Saint-Antoine, Paris
  - CHU ROUEN - Service Gastro-entérologie, Rouen
  - CHU de Saint Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No